CLINICAL TRIAL: NCT03888612
Title: A Phase 1/2, Open-label, Dose Escalation, and Cohort Expansion Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARV-110 in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Trial of ARV-110 in Patients With Metastatic Castration Resistant Prostate Cancer
Acronym: mCRPC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arvinas Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARV-110-mCRPC-101
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Metastatic
Keywords: Metastatic Prostate Cancer; Castrate-Resistant; Prostate Cancer; mCRPC; adenocarcinoma of the prostate; bavdegalutamide
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARV-110 (Experimental): Part A: Oral tablet(s), once or twice daily in 28 day cycles
  Part B: Oral tablet(s), once or twice daily in 28 day cycles
  Interventions: Drug: ARV-110

INTERVENTIONS:
Drug: ARV-110 — Part A: Daily oral dosages are predetermined by cohort review committee after the initial starting dose cohort after the first 28 days of treatment
  Part B: Daily oral dosage and schedule at a recommended Phase 2 dose based on data from Part A

SUMMARY:
Phase 1/2 dose escalation study to assess the safety and tolerability of ARV-110 in men with mCRPC who have progressed on prior approved systemic therapies for their castrate resistant disease (one of which must be enzalutamide or abiraterone).

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Patients must be male and at least 18 years of age at the time of signing the informed consent.
* Patients must present with histological, pathological, or cytological confirmed diagnosis of advanced or metastatic castration resistant adenocarcinoma of the prostate.
* Patients must have progressed on at least 2 prior approved systemic therapies for CRPC (at least one must be abiraterone or enzalutamide).
* Patients with progressive mCRPC
* Patients must have ongoing ADT with a gonadotropin releasing hormone analog or inhibitor, or orchiectomy (surgical or medical castration).

Part B:

* Patients must be male and at least 18 years of age at the time of signing the informed consent.
* Patients must present with histological, pathological, or cytological confirmed diagnosis of advanced or metastatic castration resistant adenocarcinoma of the prostate.
* Patients must have received at least one but no more than two prior second generation anti-androgen agents (e.g., enzalutamide or abiraterone) for CRPC.
* Patients must have received no more than one prior chemotherapy regimen in each of the following settings: castrate sensitive and castrate resistant prostate cancer.
* Patients must have ongoing ADT with a gonadotropin releasing hormone analog or inhibitor, or orchiectomy (surgical or medical castration).

Part B - Phase 2 Expansion Cohort Subgroup 4

* Patient has received only one prior AR second generation therapy (e.g., abiraterone or enzalutamide) either as treatment for CSPC or CRPC and no more than 1 regimen in CRPC setting.
* No prior chemotherapy

Exclusion Criteria:

Part A:

* Patients with known symptomatic brain metastases requiring steroids (above physiologic replacement doses)
* Major surgery (as defined by the Investigator) within 4 weeks of first dose of study drug.
* Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow. Palliative radiation for the alleviation of pain due to bone metastasis will be allowed during the study
* Systemic anti cancer therapy within 2 weeks of first dose of study drug (6 weeks for bicalutamide, mitomycin C, or nitrosoureas and 4 weeks for abiraterone). Patients are ineligible if they received any other type of anti cancer agent (except agents to maintain castrate status) within 2 weeks before first dose of study drug.

Part B:

* Patients with known symptomatic brain metastases requiring steroids (above physiologic replacement doses)
* Major surgery (as defined by the Investigator) within 4 weeks of first dose of study drug.
* Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow. Palliative radiation for the alleviation of pain due to bone metastasis will be allowed during the study
* Systemic anti cancer therapy within 2 weeks of first dose of study drug (6 weeks for bicalutamide, mitomycin C, or nitrosoureas and 4 weeks for abiraterone). Patients are ineligible if they received any other type of anti cancer agent (except agents to maintain castrate status) within 2 weeks before first dose of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of Dose Limiting Toxicities of ARV-110 | 28 Days
  First Cycle Dose limiting toxicities characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug
Part A: Number of Patients with Adverse Events as a measure of safety and tolerability of ARV-110 | 28 Days
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug.
Part A: Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-110 | 28 Days
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Part B: Measurement of PSA response rate per PCWG3 accessing anti-tumor activity of ARV-110 | 12 Weeks
  PSA response rate per PCWG3.
Part B: Measurement of overall RECIST response rate accessing the anti-tumor activity of ARV-110 | 12 Weeks
  Overall RECIST response rate in patients with measurable disease at baseline.
Part B: To evaluate the clinical anti-tumor activity of ARV-110 in patients with mCRPC | 12 Weeks
  To evaluate the clinical anti-tumor activity (PSA response rate per PCWG3, Overall RECIST RR, rPFS, and PFS) of ARV-110 in patients with mCRPC in different subgroups of patients with mCRPC with predefined tumor genomic and molecular profiles or based on prior therapy.

SECONDARY OUTCOMES:
Part A: Anti-tumor activity based on the overall PSA response in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the overall PSA response per PCWG3.
Part A: Anti-tumor activity based on the overall RECIST response in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the overall RECIST response rate.
Part A: Anti-tumor activity based on the progression free survival in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the time to event progression free survival.
Part A: Anti-tumor activity based on the duration of response in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the duration of response.
Part A: Anti-tumor activity based on the time to progression in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the time to progression.
Part A: Anti-tumor activity based on the overall survival in the entire study population and in the subsets of patient based on the AR mutational status of their tumor. | 12 Weeks
  The anti-tumor activity of ARV-110 will be assessed by evaluating the overall survival.
Part A: Concentration-time curve (AUC) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC).
Part A: Maximum concentration (Cmax) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter maximum concentration (Cmax).
Part A: Minimum concentration (Cmin) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter minimum concentration (Cmin).
Part A: Time to maximum concentration (Tmax) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter time to maximum concentration (Tmax)
Part B: Concentration-time curve (AUC) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter area under the concentration-time curve (AUC).
Part B: Maximum concentration (Cmax) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter maximum concentration (Cmax).
Part B: Minimum concentration (Cmin) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter minimum concentration (Cmin).
Part B: Time to maximum concentration (Tmax) for single and multiple dose of ARV-110 | 28 Days
  PK parameters will be assessed when applicable after a single dose and after multiple once and twice daily doses. Assessment of pharmacokinetic parameter time to maximum concentration (Tmax)
Part B: Duration of response | 12 Weeks
  From the date of first confirmed best overall response of CR or PR to the date of first progression per RECIST 1.1 or PCWG3, or death due to any cause without evidence of radiographic progression, whichever occurs first.
Part B: Overall survival | 12 Weeks
  Time interval from the date of first ARV-110 dose to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (54):
- United States (54):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, San Francisco, California
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Altamonte Springs, Florida
  - Clinical Trial Site, Bonita Springs, Florida
  - Clinical Trial Site, Bradenton, Florida
  - Clinical Trial Site, Brandon, Florida
  - Clinical Trial Site, Cape Coral, Florida
  - Clinical Trial Site, Clearwater, Florida
  - Clinical Trial Site, Daytona Beach, Florida
  - Clinical Trial Site, Fleming Island, Florida
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Gainesville, Florida
  - Clinical Trial Site, Largo, Florida
  - Clinical Trial Site, Lecanto, Florida
  - Clinical Trial Site, Naples, Florida
  - Clinical Trial Site, New Port Richey, Florida
  - Clinical Trial Site, Ocala, Florida
  - Clinical Trial Site, Orange City, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, Port Charlotte, Florida
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Spring Hill, Florida
  - Clinical Trial Site, St. Petersburg, Florida
  - Clinical Trial Site, Stuart, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Tavares, Florida
  - Clinical Trial Site, The Villages, Florida
  - Clinical Trial Site, Venice, Florida
  - Clinical Trial Site, Vero Beach, Florida
  - Clinical Trial Site, Wellington, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Winter Park, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Las Vegas, Nevada
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Dickson, Tennessee
  - Clinical Trial Site, Franklin, Tennessee
  - Clinical Trial Site, Gallatin, Tennessee
  - Clinical Trial Site, Hendersonville, Tennessee
  - Clinical Trial Site, Hermitage, Tennessee
  - Clinical Trial Site, Lebanon, Tennessee
  - Clinical Trial Site, Murfreesboro, Tennessee
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Shelbyville, Tennessee
  - Clinical Trial Site, Smyrna, Tennessee
  - Clinical Trial Site, Salt Lake City, Utah
  - Clinical Trial Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Snyder LB, Neklesa TK, Willard RR, Gordon DA, Pizzano J, Vitale N, Robling K, Dorso MA, Moghrabi W, Landrette S, Gedrich R, Lee SH, Taylor ICA, Houston JG. Preclinical Evaluation of Bavdegalutamide (ARV-110), a Novel PROteolysis TArgeting Chimera Androgen Receptor Degrader. Mol Cancer Ther. 2025 Apr 2;24(4):511-522. doi: 10.1158/1535-7163.MCT-23-0655. PMID 39670468